CLINICAL TRIAL: NCT02069210
Title: The Immunomodulation Effect of Blood Transfusion in Operative Spine Surgery Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Collaborators: Wolf-Schleinzer-Stiftung (Unknown)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associated Professor, Mahidol University
Other Study IDs: SI 1
Record Dates: First submitted 2014-02-17; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Infection After Transfusion
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood transfusion: Patients receive blood transfusion during operation
  Interventions: Other: Blood transfusion

INTERVENTIONS:
Other: Blood transfusion — Intraoperative blood transfusion

SUMMARY:
The purpose of this study is to investigate the effect of transfusion of allogeneic (homologous) red cells on the immunologic parameters such as T-cells as well as natural killer cell count/function, various interleukins, TNF alpha and other immunologic relevant parameters on postoperative day 1,3 and 5-7 in patients undergoing spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 - < 60 years
* Patients underwent elective spine surgery
* ASA classification 1-3

Exclusion Criteria:

* Patients who have the concomitant condition
* Cancer
* History of heart disease including, heart failure, coronary artery disease, hypertension treated with more than one medicament.
* Serum creatinine > 1.5 mg/dL
* Stroke, neurologic and mental deficits, epilepsy
* General or local infection (site of surgery),
* Coagulation disorders.
* Intraoperative massive bleeding
* Infection of the spine
* Rheumatoid arthritis
* Patients who had either of the following drug (aspirin, methotrexate, cyclosporine, qualaquin)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients underwent elective spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Immunologic parameters | 7 days
  Blood level of the following parameters on preoperative, postoperative day 1, 3, 5-7.
  1. IL-1beta, IL-1ra, IL-2, IL-4, IL-5, IL-6, Il-7, IL-8, Il-9, Il-10, Il-12, Il-13, IL-15, Il-17,basic FGF (Fibroblast growth factors).
  2. Cell Analytics - (mononuclear) T-Cells incl. killer cells, CD2, CD3, CD4, CD8, CD25, CD30, CD19, CD20, CD138, CD56, CD56, CD303, CD304, NK cytotoxicity (non-radioisotope), CTL cytotoxicity (non-radioisotope), T cell proliferation, B cell, T cell.

SECONDARY OUTCOMES:
To determine the effect of red cell transfusion on clinical relevant outcome parameters, such as myocardial infarction, infection rate, and length of hospital stay. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Study Director — Department of Anesthesiology, Faculty of medicine Siriraj Hospital, Mahidol University
Locations (1):
- Sirilak Suksompong, Bangkok, Thailand